CLINICAL TRIAL: NCT01868594
Title: Multicentre Double-blind Placebo-controlled Parallel-group Randomized Clinical Trial of Efficacy and Safety of Subetta in the Combined Treatment of Patients With Type I Diabetes Mellitus
Brief Title: Clinical Trial of Efficacy and Safety of Subetta in the Combined Treatment of Patients With Type I Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MMH-SU-003
Record Dates: First submitted 2013-05-27; First posted 2013-06-04 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Type I Diabetes Mellitus
Keywords: Combined treatment of patients with type I diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — subetta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subetta group (Experimental): Patients with poor glycemic control (HbA1c=7.0-10.0%) in basal-bolus insulin regimen with a stable basal insulin dose (permissible fluctuations are ±10%) during the previous 3 months are included
  Interventions: Drug: Subetta
- Placebo group (Placebo Comparator): Patients with poor glycemic control (HbA1c=7.0-10.0%) in basal-bolus insulin regimen with a stable basal insulin dose (permissible fluctuations are ±10%) during the previous 3 months are included.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Subetta — Each Subetta tablet contains a mixture of affinity purified polyclonal antibodies to β-subunit of the rINS (6 mg) and antibodies to eNOS (6 mg) in released-active form produced by the patented technology in accordance with the applicable European Pharmacopeia requirements.
  Standard therapy of type I diabetes mellitus + Subetta (1 tablet 4 times a day) for 36 weeks.
  Subetta: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Arms: Subetta group
Drug: Placebo — Placebo (identical to Subetta in shape and taste tablet containing exсipients). Standard therapy of type I diabetes mellitus + Placebo (1 tablet 4 times a day) for 36 weeks.
  Placebo: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Arms: Placebo group

SUMMARY:
The purpose of this study is:

* to assess clinical efficacy of Subetta in the combined treatment of type I diabetes mellitus;
* to assess safety of Subetta in the combined treatment of type I diabetes mellitus.

DETAILED DESCRIPTION:
Patients with type I diabetes mellitus are included in the trial. It is concerned those patients, who by the time of the trial receive basal bolus insulin therapy of type I diabetes mellitus, including basal insulin (using long acting medications) and prandial insulin (short and ultra short acting medications), and with poor glycemic control (HbA1c=7.0-10.0%). For patients, which will be included in the trial (mainly middle aged patients without severe complications of diabetes), HbA1c>7.0% is the marker showing that optimal individual goal of glycemic control is not achieved.

HbA1c, fasting plasma glucose, microalbuminuria, estimated glomerular filtration rate, ophthalmoscopy, blood pressure measurement, patient self-monitoring of blood glucose, frequency of hypoglycemia, endocrinologist examination were performed within screening period. Patients without severe diabetes complications are randomized in 2 groups.

If a patient meets inclusion criteria and does not show exclusion criteria he/she is randomized in one of 2 groups: Group 1 - patients receiving standard type I diabetes mellitus therapy + Subetta at a dose of 1 tablet 4 times a day; Group 2 - the group receiving standard type I diabetes mellitus therapy + Placebo under the regimen used for Subetta. The invented names of the drugs containing basal and prandial (meal) insulin should be unchanged for each patient during the whole trial.

All patients will receive glucometers and the appropriate glucose test strips, so they could self monitor blood glucose and register this data in their diaries.

The trial duration is 38 weeks; the main stages of the trial are conducted during screening, then in 4 weeks (Visit 2), in 12 weeks (Visit 3), in 24 weeks (Visit 4) and in 36 weeks (Visit 5). In 1 week after randomization and the onset of the trial therapy and between the visits to the study site (on weeks 8±1, 18±1 and 30±1) an investigator collects data on patient's health and complaints (phone visits) to decide whether it is necessary to arrange unplanned visit to the site.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed type I diabetes mellitus (according to WHO criteria, 1999 - 2006).
2. Disease duration no less than 6 months.
3. Patient's age from 18 to 65 years inclusive.
4. Level of glycosylated hemoglobin 7.0- 10.0 %.
5. Glomerular filtration rate ≥ 60 ml/ min/1.73m^2.
6. Stable dose of basal insulin for the last 3 months. (Permissible fluctuations are ±10%.)
7. Usage of contraceptive methods by both gender patients of reproductive age during the trial and within 30 days after ending the participation in the trial.
8. Availability of signed patient information sheet (Informed Consent form) for participation in the clinical trial.

Exclusion Criteria:

1. Acute diabetes mellitus complications for 3 months prior to inclusion in the trial (diabetic ketoacidosis, hyperosmolar hyperglycemic state, lacticemia, severe hypoglycemia and hypoglycemic coma).
2. Diabetic retinopathy, preproliferative, proliferative or terminal stages (based on the results of oculist examination during screening period or 6 months prior to the trial).
3. Diabetic nephropathy, proteinuria stage, chronic kidney disease on 3, 4 or 5 stage.
4. Diabetic microangiopathy:

   * ishemic heart disease (medical history of a sudden coronary death with successful reanimation, medical history of myocardial infarction, stable exertional angina III or IV FC; unstable angina; post-infarction cardiosclerosis; chronic heart failure III or IV FC);
   * cerebrovascular diseases (medical history of acute cerebrovascular accident; progressive vascular leukoencephalopathy; vascular dementia);
   * chronic obliterative peripheral vascular diseases (clinically significant);
   * diabetic neuroosteoarthropathy;
   * diabetic foot (clinically significant).
5. Heart rhythm disorder:

   * II-III atrioventricular block;
   * sick sinus syndrome;
   * long QT interval syndrome;
   * complete left bundle branch block;
   * block of 2/3 bundle branches;
   * WPW syndrome;
   * ventricular arrhythmia of III grade according Laun-Wolf;
   * paroxysmal supraventricular tachycardia;
   * paroxysmal/recurrent ventricular tachycardia;
   * atrial flutter and fibrillation;
   * ventricular flutter and fibrillation;
   * heart pacemaker implant.
6. Uncontrolled arterial hypertension characterized by the following blood tension values: systolic blood pressure over 160 mm Hg and/or diastolic blood pressure over 100 mm Hg.
7. Severe concomitant pathology including clinically significant cardiovascular diseases of III - IV functional class (according to New York Heart Association classification, 1964), nervous and endocrine system diseases, including morbid obesity (body mass index≥40.0 kg/m2), renal insufficiency, liver failure.
8. Medical history of pancreatectomy or transplantation of pancreatic/islet cells.
9. Medical history of renal transplantation.
10. Malignant neoplasms/suspected malignant neoplasms.
11. Exacerbations or decompensation of chronic diseases affecting a patient's ability to participate in the clinical trial.
12. Level of fasting triglycerides >5.64 mmol/L.
13. Medical history of bariatric surgical operations.
14. Medical history of polyvalent allergy.
15. Allergy/ intolerance to any of the components of medications used in the treatment.
16. Intake of medicines listed in the section "Prohibited concomitant treatment" for 3 months prior to the inclusion in the trial.
17. Pregnancy, breast-feeding.
18. Drug addiction, alcohol usage in the amount exceeding 2 units of alcohol per day.
19. Mental disorders of a patient.
20. Night work.
21. Participation in other clinical trials in the course of 3 months prior to the inclusion in the trial.
22. Patients, who from the investigator's point of view, will fail to comply with the observation requirements of the trial or with the intake regimen of the investigated medicines.
23. Other factors impeding patient's participation in the trial (for example, planned business trips or journeys).
24. Patient is related to the research personnel of the investigative site, who are directly involved in the trial or are the immediate relative of the researcher. The immediate relative includes husband/wife, parents, children or brothers (or sisters), regardless of whether they are natural or adopted.
25. Patient works for OOO "NPF "Materia Medica Holding" (i.e. is the company's employee, temporary contract worker or appointed official responsible for the carrying out the research) or the immediate relative.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- Russia (15):
  - State Healthcare Institution of Moscow "Central research institute of gastroenterology" of Department of health care of Moscow, Moscow
  - State Educational Institution of Higher Professional Education "Moscow State Medical Academy named after I.M. Sechenov", Moscow
  - Nonstate Health Care Institution "Central Clinical Hospital №2 named after N.A. Semashko of Public Limited Company "Russian Railways", Moscow
  - Municipal budgetary authority "Khimki Central Clinical Hospital", Moscow Region
  - The State Budgetary Institution of Health Care of the Nizhny Novgorod Region "City clinical hospital No. 10 ", Nizhny Novgorod
  - Nizhny Novgorod regional State Budgetary Health Institution " Nizhny Novgorod regional Clinical Hospital named after N.A. Semashko ", Nizhny Novgorod
  - State Budgetary Educational Institution of High Professional Training "Rostov State Medical University" of Ministry of Health of Russian Federation, Department of Endocrinology, Rostov-on-Don
  - Private company "Polyclinic Complex", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "City Polyclinic №6", Saint Petersburg
  - St. Petersburg State Budgetary Health Care Institution "Saint Venerable Martyr Elizaveta Municipal Hospital", Saint Petersburg
  - State Budgetary Educational Institution of High Professional Training "St. Petersburg State Medical University named after academician I.P. Pavlov" of Ministry of Health of Russian Federation, Therapy Faculty Board, Saint Petersburg
  - St. Petersburg Sate Budgetary Institution "Consultative-Diagnostic Polyclinic №1 of Coastal Area", Saint Petersburg
  - Co.Ltd " Diabet Center", Samara
  - Independent Health Care Institution of Voronezh Region "Voronezh Regional Clinical Consultative-Diagnostic Center", Voronezh
  - State Budgetary Health Care Institution of Yaroslavl Region "Regional Сlinical Hospital", Yaroslavl

REFERENCES:
- [Derived] Mkrtumyan A, Romantsova T, Vorobiev S, Volkova A, Vorokhobina N, Tarasov S, Putilovskiy M, Andrianova E, Epstein O. Efficacy and safety of Subetta add-on therapy in type 1 diabetes mellitus: The results of a multicenter, double-blind, placebo-controlled, randomized clinical trial. Diabetes Res Clin Pract. 2018 Aug;142:1-9. doi: 10.1016/j.diabres.2018.04.044. Epub 2018 May 26. PMID 29807102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled patients using intensive insulin regimen (Short-acting and Long-acting human insulins) with type 1 diabetes who were not meeting glycemic control (HbA1c>7.0%). Eligible patients were assessed by endocrinologists. The study was performed in 15 medical institutions in Russia from May 2013 to October 2015.
Pre-assignment Details: Selection procedures were carried out after participant enrollment to determine whether the patient could participate in the study in accordance with the inclusion/exclusion criteria.
  Of the 200 patients enrolled, 49 did not meet inclusion criteria after screening procedures, they were not randomized
Groups:
- Subetta: Short-acting and Long-acting human insulins + Subetta (1 tablet 4 times a day). Subetta: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Subetta: Efficacy and Safety of Subetta in the combined treatment of patients with type I diabetes mellitus
- Placebo: Short-acting and Long-acting human insulins + Placebo (1 tablet 4 times a day). Placebo: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Placebo
Period: Overall Study
Arm/Group | Subetta | Placebo
Started | 76 | 75
Completed | 72 | 72
Not Completed | 4 | 3
Not completed — Do not meet inclusion criteria | 4 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-Treat set
Groups:
- Total: Total of all reporting groups
Arm/Group | Subetta | Placebo | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.2 (9.6) | 35.0 (10.4) | 36.1 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 36 | 70
  Male | 38 | 36 | 74
Weight [Mean (Standard Deviation); unit: kilogram] | 77.7 (15.2) | 74.4 (13.5) | 76.0 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Mean Value of HbA1c
Description: The HbA1C test was performed using a method that is certified by the National Glycohemoglobin Standardization Program (NGSP) (www.ngsp.org) and standardized or traceable to the Diabetes Control and Complications Trial (DCCT) reference assay.
Time Frame: baseline and 12, 24 and 36 weeks of the treatment
Population: Intention-to-Treat set
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 72 | 72
percentage of HbA1c
  12 weeks | -0.71 (0.91) | -0.49 (1.02)
  24 weeks | -0.66 (0.94) | -0.27 (1.13)
  36 weeks | -0.59 (0.99) | -0.20 (1.14)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.019, Mixed Models Analysis — The p-value associated with "treatment" factor of changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

2. Secondary Outcome: Change in Fasting Plasma Glucose (Based on the Data of Biochemical Analysis)
Time Frame: baseline and 4, 12, 24 and 36 weeks of the treatment
Population: Intention-to-Treat set
Measure: Mean (Standard Deviation); unit: mmol / l
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 72 | 72
mmol / l
  4 weeks | -0.5 (5.1) | 0.3 (4.6)
  12 weeks | -0.2 (4.8) | 0.8 (4.9)
  24 weeks | -0.7 (4.9) | 0.7 (5.4)
  36 weeks | -0.8 (4.8) | 1.1 (5.4)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.0432, Mixed Models Analysis — The p-value associated with "treatment" factor of changes from baseline to Week 4, 12, 24 and 36 endpoint between Subetta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

3. Secondary Outcome: Change in Average Daily Blood Glucose From a 7-point Patient Self-monitoring of Blood Glucose (SMBG)
Description: A 7-point patient self-monitoring of blood glucose (SMBG):
  three measurements of blood glucose before the meal; three measurements of postprandial blood glucose (1-2 h after the start of the meal) and one measurement at 3:00 a.m.
Time Frame: baseline and 4, 8, 12, 18, 24, 30 and 36 weeks of the treatment
Population: Intention-to-Treat. 2 patients (1 in Subetta group and 1 in Placebo group) was excluded from the analysis due to lake of diaries
Measure: Mean (Standard Deviation); unit: mmol / l
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 71 | 71
mmol / l
  4 weeks | -0.1 (1.4) | 0.1 (1.8)
  8 weeks | -0.2 (1.7) | -0.1 (2.0)
  12 weeks | -0.2 (1.6) | -0.2 (2.0)
  18 weeks | -0.1 (2.2) | -0.1 (1.9)
  24 weeks | -0.3 (1.7) | 0.0 (2.0)
  30 weeks | 0.0 (1.8) | -0.1 (1.8)
  36 weeks | -0.1 (1.9) | 0.0 (2.0)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.7344, Mixed Models Analysis — The p-value associated with "treatment" factor of changes from baseline to Week 4, 8, 12, 18, 24, 30 and 36 endpoint between Subetta and Placebo treatment groups. Model includes treatment, visit and treatment*visit interaction

4. Secondary Outcome: Changes in Lipids (Concentrations of Plasma Total Cholesterol, HDL Cholesterol, LDL Cholesterol and Triglycerides)
Description: Blood samples (for measurement of fasting plasma glucose, concentrations of plasma total cholesterol, HDL cholesterol, LDL cholesterol and triglycerides) are taken under standard conditions: after night break in food taking (at least 12 hours) and prior to administering of insulin morning dose (prandial), prior to any morning medicines intake (including the study drug and permitted concomitant therapy).
Time Frame: baseline and 12, 24 and 36 weeks of the treatment
Population: Intention-to-Treat set
Measure: Mean (Standard Deviation); unit: mmol / l
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 72 | 72
mmol / l
  Total cholesterol (12 weeks) | 0.2 (1.0) | 0.2 (0.9)
  Total cholesterol (24 weeks) | 0.1 (1.1) | 0.4 (1.2)
  Total cholesterol (36 weeks) | 0.2 (1.0) | 0.3 (1.2)
  HDL cholesterol (12 weeks) | 0.1 (0.3) | 0.0 (0.3)
  HDL cholesterol (24 weeks) | 0.0 (0.3) | 0.0 (0.3)
  HDL cholesterol (36 weeks) | 0.1 (0.3) | 0.0 (0.3)
  LDL cholesterol (12 weeks) | 0.2 (0.8) | 0.2 (0.6)
  LDL cholesterol (24 weeks) | 0.0 (0.9) | 0.3 (0.9)
  LDL cholesterol (36 weeks) | 0.1 (0.8) | 0.3 (0.9)
  Triglycerides (12 weeks) | -0.1 (0.6) | 0.1 (0.8)
  Triglycerides (24 weeks) | -0.1 (0.6) | 0.0 (0.6)
  Triglycerides (36 weeks) | -0.1 (0.6) | 0.1 (0.8)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Analysis of Total cholesterol changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.2780, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Subetta vs Placebo; Analysis of HDL cholesterol changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.8114, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Subetta vs Placebo; Analysis of LDL cholesterol changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.1619, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Subetta vs Placebo; Analysis of Triglycerides changes from baseline to Week 12, 24 and 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.0764, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

5. Secondary Outcome: Changes in Dosage of Insulin (Basal, Prandial and Total Daily Dose Insulin Measured in IU)
Description: Insulin dose should be corrected by a patient on a daily basis taking into consideration data on blood glucose self- monitoring during a day and amount of food carbohydrates. Physician can correct insulin dose based on the same data.
Time Frame: baseline and 36 weeks of the treatment
Population: Intention-to-Treat set
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 72 | 72
IU
  Basal insulin (36 weeks) | 0.4 (2.4) | 0.9 (2.9)
  Prandial insulin (36 weeks) | -1.6 (6.9) | -0.9 (4.5)
  Total daily dose insulin (36 weeks) | -1.2 (8.3) | 0.0 (6.2)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Analysis of basal insulin changes from baseline to Week 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.3107, t-test, 2 sided — The p-value associated with comparison of changes from baseline to Week 36 endpoint between Subetta and Placebo treatment groups
Statistical Analysis 2: Comparison: Subetta vs Placebo; Analysis of prandial insulin changes from baseline to Week 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.5236, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Subetta vs Placebo; Analysis of total daily dose insulin changes from baseline to Week 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.3847, t-test, 2 sided — [p-value comment as in outcome 5, analysis 1]

6. Secondary Outcome: Changes in Dosage of Total Insulin Measured in IU/kg of Body Weight
Description: as for outcome 5
Time Frame: baseline and 36 weeks of the treatment
Population: Intention-to-Treat set
Measure: Mean (Standard Deviation); unit: IU/kg
Groups:
- Subetta: Standard therapy of type I diabetes mellitus + Subetta (1 tablet 4 times a day).
  Subetta: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Subetta: Efficacy and Safety of Subetta in the combined treatment of patients with type I diabetes mellitus
- Placebo: Standard therapy of type I diabetes mellitus + Placebo (1 tablet 4 times a day).
  Placebo: oral administration, per 1 intake - 1 tablet (keep in the mouth until complete dissolution, not at mealtime).
  Placebo
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 72 | 72
IU/kg | -0.02 (0.09) | -0.01 (0.08)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Test type: Superiority; p = 0.6716, t-test, 2 sided

7. Secondary Outcome: Satisfaction of Diabetes Treatment Based on Diabetes Treatment Satisfaction Questionnaire Data
Description: The Diabetes Treatment Satisfaction Questionnaire allows to assess the degree of satisfaction with treatment for diabetes and its complications - retinopathy and nephropathy, how patients' satisfaction and perceived hyper- and hypoglycemia have changed compared to the initial period (before the treatment).
  The Diabetes Treatment Satisfaction Questionnaire contains six items scored on 7-point scales from +3 (equals "very satisfied") to -3 (equals "very dissatisfied"), with 0 (equals "no change"). These are summed to produce a total Treatment Satisfaction score. Two questions concerning "Perceived Hyperglycaemia" and "Perceived Hypoglycaemia" respectively, are calculated separately. According to these two items, low scores represent good perceived blood glucose control (+3 means "most of the time" of Hyperglycaemia or Hypoglycaemia whereas -3 means "none of the time" of Hyperglycaemia or Hypoglycaemia).
Time Frame: 36 weeks of the treatment
Population: Intention-to-Treat set. 6 patients (1 in the Subetta group and 5 in the Placebo group) was excluded from the analysis due to lake of questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subetta | Placebo
Number analyzed (Participants) | 71 | 67
score on a scale
  Satisfaction | 9.7 (6.6) | 8.4 (6.5)
  Hyperglycemia | -0.7 (1.5) | -0.6 (1.6)
  Hypoglycemia | -0.4 (1.6) | -0.6 (1.4)
Statistical Analysis 1: Comparison: Subetta vs Placebo; Analysis of total Treatment Satisfaction score at Week 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.2484, t-test, 2 sided — The p-value associated with comparison of Week 36 endpoint between Subetta and Placebo treatment groups
Statistical Analysis 2: Comparison: Subetta vs Placebo; Analysis of "Perceived Hyperglycaemia" question at Week 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.7610, t-test, 2 sided — The p-value associated with comparison of Week 36 endpoint between Subetta and Placebo treatment groups
Statistical Analysis 3: Comparison: Subetta vs Placebo; Analysis of "Perceived Hypoglycemia" question at Week 36 endpoint between Subetta and Placebo treatment groups; Test type: Superiority; p = 0.3714, t-test, 2 sided — The p-value associated with comparison of Week 36 endpoint between Subetta and Placebo treatment groups

ADVERSE EVENTS:
Time Frame: Adverse/Serious adverse events were registered during 36 weeks of therapy and 30 days after the end of therapy.
Description: Adverse/Serious adverse events were registered in patients of the Full Analysis Set (n=151, Safety Population)
Arm/Group | Subetta | Placebo
Serious Adverse Events (participants affected / at risk) | 2/76 | 3/75
Other Adverse Events (participants affected / at risk) | 16/76 | 18/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subetta (N=76) | Placebo (N=75)
Hypertension arterial (Vascular disorders) | 1 | 0
Fracture of humerus (Injury, poisoning and procedural complications) | 1 | 0
Parotid abscess (Infections and infestations) | 0 | 1
Chronic venous insufficiency (Vascular disorders) | 0 | 1
Varicose veins of lower extremities (Vascular disorders) | 0 | 1
Type I diabetes mellitus with ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subetta (N=76) | Placebo (N=75)
Inflammation of inguinal lymphonodus on the right (Blood and lymphatic system disorders) | 0 | 1
Goiter (Endocrine disorders) | 1 | 0
Subclinical hypothyreoidism (Endocrine disorders) | 1 | 0
Bacterial food poisoning (Gastrointestinal disorders) | 1 | 0
Heartburn (Gastrointestinal disorders) | 1 | 0 — exacerbation of chronic gastritis
Epigastric pain (Gastrointestinal disorders) | 0 | 1
Dentalgia (Gastrointestinal disorders) | 0 | 1
Increase in body temperature to 38.5 C (General disorders) | 0 | 2
Increase in body temperature up to 38.2 С (General disorders) | 0 | 1
Diabetic hepatosis (Hepatobiliary disorders) | 1 | 0
Allergic reactions (Immune system disorders) | 0 | 1
Angina (Infections and infestations) | 0 | 1
Acute respiratory viral infection (Infections and infestations) | 5 | 3
Acute respiratory disease (Infections and infestations) | 0 | 3
Acute bronchitis (Infections and infestations) | 0 | 3
Parodontosis (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Contusion of the hand (Injury, poisoning and procedural complications) | 0 | 1
Palpitations (Investigations) | 1 | 0
Increased blood pressure to 150/90 mm Hg, headache, nausea (Investigations) | 0 | 1
Increased body temperature (Investigations) | 0 | 1
Fasting hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 2
Pain in the shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1
Heavy legs (Musculoskeletal and connective tissue disorders) | 1 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 0
Cervicalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Headache (Nervous system disorders) | 5 | 2
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Increased blood pressure (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes